





| SOP Plan d'analy | se statistique | |
|-------------------------|----------------|----------------|
| SOP CRC-CHUV DM201 AN01 | | |
| 005 4050 | | Version : V01 |
| Création : | Yolanda Mülle | r / 29.11.2018 |
| Révision : | -1 | 4 6 |
| Approbation: | IL, NS | |

# STATISTICAL ANALYSIS PLAN

Protocol title:

Efficacy of an Active Geriatric Evaluation for geriatric syndromes (AGE

tool) to prevent functional decline in elderly patients in family

medicine: a pragmatic cluster randomized trial

Protocol number:

ClinicalTrials.gov NCT02618291; CER-VD 2016-00422

Protocol version and date: Version 8, 01/05/2018

SAP author:

Yolanda Müller Chabloz

SAP version:

v1, 29.11.2018

SAP Revision:

SAP implementation : Yolanda Müller Chabloz, Isabella Locatelli

Reference person : Yolanda Müller Chabloz

## CONFIDENTIEL

Le plan d'analyses statistiques doit être préparé par le chercheur et le statisticien, afin de décider de la meilleure approche pour répondre aux objectifs de l'étude. Ainsi, le SAP doit être rédigé par le(s) chercheur(s) et par le statisticien : le statisticien responsable doit écrire le SAP, ou le passer en revue si l'investigateur fournit un SAP complet. Les auteurs du SAP sont responsables de s'assurer que le SAP soit produit en suivant les spécifications correctes de l'étude et de le faire parvenir pour révision à l'investigateur







Programme AGE
Centre de recherche et développement
PMU | Policlinique médicale universitaire
Rue du Bugnon 44 | BU44 04-2316

1011 Lausanne | Suisse Tél 021 314 32 94 ou 079 556 11 48

| SOP Plan d'ana | lyse statistique | 9 |
|----------------|------------------|--------------------|
| SOP CRC-CH | HUV DM201 | AN01 |
| SOP AGE3 DM | AN01 | Version : V01 |
| Création : | Yolanda M | üller / 29.11.2018 |
| Révision : | | |
| Approbation: | IL, NS | |

Version 1, 29.11.2018

# **Approbation:**

Approved by:

Name:.

Dr Yolanda Müller Chabloz

Study coordinator

Nom:.

Dr Isabella Locatelli

Study statistician

Nom:.

Prof Nicolas Senn

Principal investigator

Date

Date

18,1.20

Date 14.12

3







| SOP Plan d'ana | ılyse statistiqı | ue |
|----------------|------------------|---------------------|
| SOP CRC-CI | HUV DM20 | 1 AN01 |
| Création : | Yolanda N | Müller / 29.11.2018 |
| Révision : | | |
| Approbation: | IL, NS | |

# **Table of content**

# Table des matières

| Stat | istical <i>F</i> | Analysis Plan | |
|---|---|---|---|
| Abb | reviatio | ons | Ę |
| 1. | | y objectives | |
| | 1.1. | Overall Objective | |
| | 1.2. | Primary Objective | |
| | 1.3. | Secondary Objectives | |
| | 1.4. | Safety Objectives | |
| 2. | Rese | earch questions and hypotheses | |
| | 2.1. 8 | Efficacy : | 7 |
| 3. | Modi | fications of study objectives during the study | 11 |
| 4. | | y design | |
| 5. | | ılation - sampling | |
| 6. | | sary of study variables | |
| 7. | Statis | stical analyses | 33 |
| | 7.1 | Intermediate analyses | |
| | 7.2 | Final data analysis | |
| 8. | Refe | rences | |







SOP Plan d'analyse statistique SOP CRC-CHUV DM201 AN01

Approbation:

Programme AGE

Centre de recherche et développement PMU | Policlinique médicale universitaire

Rue du Bugnon 44 | BU44 04-2316

1011 Lausanne | Suisse

Tél 021 314 32 94 ou 079 556 11 48

Email Davi ano@haanid ah

Version: V01 SOP AGE3 DM AN01 Yolanda Müller / 29.11.2018 Création: Révision:

IL, NS

## ABBREVIATIONS

Activities of Daily Living ADL

Adverse Event ΑE

Active Geriatric Evaluation AGE **Brief Assessment Tool** BAT

Commission d'Ethique de la Recherche sur l'être humain du canton de

**CER VD** Vaud

Centre de Recherche Clinique CRC

Case Report Form **CRF** 

Electronic Case Report Form eCRF

Common terminology criteria for adverse events CTCAE

Family Practitioner FP Good Clinical Practice **GCP** Null hypothesis Но

Alternative hypothesis H1

Instrumental activities of daily living IADL

Interquartile range **IQR** Intention to treat ITT

Potentially Inappropriate Prescription PIM

Severe Adverse Event SAE Statistical Analysis Plan SAP

Standard Operating Procedure SOP

WHO quality of life score for the elderly WHOQOL-OLD







| SOP Plan d'ana | ılyse statistiqu | ıe |
|------------------------------|------------------|---------------------|
| SOP CRC-CI | HUV DM20 | 1 AN01 |
| SOP AGE3 DM AN01 Version : V | | Version : V01 |
| Création : | Yolanda M | lüller / 29.11.2018 |
| Révision : | | |
| Approbation: | IL, NS | |

## 1. STUDY OBJECTIVES

## 1.1. Overall Objective

The aim of the project is to determine whether an active geriatric evaluation performed in family medicine, combining a brief assessment tool (BAT) for the early diagnosis of geriatric syndromes with a structured diagnostic and management strategy (AGE tool), impacts on the functional decline and quality of life of elderly patients.

## 1.2. Primary Objective

The primary objective of this project are to determine whether the AGE tool used in family medicine:

1. reduces the functional decline of elderly patients.

## 1.3. Secondary Objectives

The secondary objectives of this project are to determine if the AGE tool used in family medicine:

- 2. improves the quality of life of elderly patients.
- 3. reduces the incidence of hospital admissions
- 4. reduces the incidence of institutionalizations
- 5. reduces the incidence of emergency visits
- 6. impacts on the number of FP outpatient visits
- 7. improves the processes of care (diagnoses and management) of elderly patients
- 8. is acceptable and feasible for patients and family practitioners

## 1.4. Safety Objectives

The **safety objective** of this project is to determine if the AGE tool administered in family medicine impacts the quality of life, hospitalization and death rate of elderly patients.







| SOP Plan d'analys | se statistique | |
|-------------------|-----------------------------|---------------|
| SOP CRC-CHU | JV DM201 | AN01 |
| | | Version : V01 |
| Création : | Yolanda Müller / 29.11.2018 | |
| Révision : | | |
| Approbation: | IL, NS | |

# RESEARCH QUESTIONS AND HYPOTHESES

## 2.1. Efficacy:

The AGE tool used in family medicine reduces the functional decline of elderly patients.

The null hypothesis is that there is no difference in the proportion of patients having lost at least one IADL after 2 years of follow-up after 2 years of follow-up, between elderly patients followed by a family practitioner using the AGE assessment and management tool and elderly patients followed in usual care.

The alternative hypothesis is that there will be a difference of at least 15% in the proportion of patients having lost at least one IADL after 2 years of follow-up, between elderly patients followed by a family practitioner using the AGE assessment and management tool, and elderly patients followed in usual care. We assume that 25% are expected to lose at least one IADL after 2 years without intervention.

Hypothesis 1.2:

The null hypothesis is that there is no difference in in the proportion of patients having lost at least one ADL after 2 years of follow-up between elderly patients followed by a family practitioner using the AGE assessment and management tool and elderly patients followed in usual care.

The alternative hypothesis is that there will be a difference of at least 15% in the proportion of patients having lost at least one ADL after 2 years of follow-up, between elderly patients followed by a family practitioner using the AGE assessment and management tool and elderly patients followed in usual care.

Hypothesis 1.3:

The null hypothesis is that there is no difference in the proportion of patients having lost at least one ADL of the combined IADL and ADL after 2 years of follow-up between elderly patients followed by a family practitioner using the AGE assessment and management tool and elderly patients followed in usual care.

The alternative hypothesis is that there will be a difference of at least 15% in the proportion of patients having lost at least one ADL of the combined IADL and ADL after 2 years of follow-up, between elderly patients followed by a family practitioner using the AGE assessment and management tool and elderly patients followed in usual care.

2. The AGE tool used in family medicine improves the quality of life of elderly patients.

Hypothesis 2.1:

The null hypothesis is that there is no difference in in the evolution of the total transformed scale of theWHOQOL-OLD score after 2 years of follow-up between elderly patients followed by a family practitioner using the AGE assessment and management tool and elderly patients followed in usual care.

The alternative hypothesis is that there will be a difference in the evolution of the standardised in total transformed scale of the WHOQOL-OLD score (0 to 100) after 2 years of follow-up, between elderly patients followed by a family practitioner using the AGE assessment and management tool and elderly patients followed in usual care.







| SOP Plan d'ana | llyse statistiq | lue |
|----------------|-----------------|---------------------|
| SOP CRC-CI | HUV DM20 | 01 AN01 |
| Création : | Yolanda | Müller / 29.11.2018 |
| Révision : | | |
| Approbation: | IL, NS | |

#### Hypothesis 2.2:

The null hypothesis is that there are no differences in all facets of the WHOQOL-OLD transformed total score after 2 years of follow-up between elderly patients followed by a family practitioner using the AGE assessment and management tool and elderly patients followed in usual care.

The alternative hypothesis is that there will be a difference on a transformed total score scale of 0 to 100) in at least one of the six facets of the WHOQOL-OLD score after 2 years of follow-up, between elderly patients followed by a family practitioner using the AGE assessment and management tool and elderly patients followed in usual care.

3. The AGE tool used in family medicine reduces the incidence of hospital admissions Hypothesis 3.1:

The null hypothesis is that there is no difference in the admission rate (number of admission per person-year) between patients of intervention and control arm

The alternative hypothesis is that there will be a relative difference of at least 10% in the admission rate (number of admission per person-year) between patients of intervention and control arm

4. The AGE tool used in family medicine reduces the incidence of institutionalizations Hypothesis 4.1:

The null hypothesis is that there is no difference in the institutionalization rate (number of institutionalization per person-year) between patients of intervention and control arm

The alternative hypothesis is that there will be a relative difference of at least 10% in the institutionalization rate (number of institutionalization per person-year) between patients of intervention and control arm

## Hypothesis 4.2:

The null hypothesis is that there is no difference in the time to institutionalization between patients of intervention and control arm

The alternative hypothesis is that there will be a difference in the time to institutionalization between patients of intervention and control arm

5. The AGE tool used in family medicine reduces the incidence of emergency visits Hypothesis 5.1:

The null hypothesis is that there is no difference in the emergency visit rate (number of emergency visit per person-year) between patients of intervention and control arm

The alternative hypothesis is that there will be a relative difference of at least 10% in the emergency visit rate (number of emergency visit per person-year) between patients of intervention and control arm

6. The AGE tool used in family medicine impacts on the number of FP outpatient visits Hypothesis 6.1:

The null hypothesis is that there is no difference in the consultation rate (number of FP consultation per person-year) between patients of intervention and control arm







| SOP Plan d'analy | se statistique | |
|------------------|-----------------------------|---------------|
| SOP CRC-CH | JV DM201 A | AN01 |
| SOP AGE3 DM A | N01 | Version : V01 |
| Création : | Yolanda Müller / 29.11.2018 | |
| Révision : | | |
| Approbation: | IL, NS | |

The alternative hypothesis is that there will be a difference of at least 10% in the consultation rate (number of FP consultation per person-year) between patients of intervention and control arm

7. The AGE tool used in family medicine improves the processes of care (diagnoses and management) of elderly patients

## Hypothesis 7.1:

Use of the AGE tool increases the number of chronic conditions diagnosed, in particular for diagnoses specifically relevant in the context of geriatric syndromes

## Hypothesis 7.2:

Use of the AGE tool increases the number of patients referred to a specialist

#### Hypothesis 7.3:

Use of the AGE tool enhances clinical assessment of patients

## Hypothesis 7.4:

Use of the AGE tool enhances communication between FPs and home-based care

## Hypothesis 7.5:

Use of the AGE tool enhances communication between FPs and patient families

#### Hypothesis 7.6:

Use of the AGE tool limits polymedication

## Hypothesis 7.6:

Use of the AGE tool limits the number of potentially inappropriate medications

The changes in these processes of care will be described by arm, without a formal predefined hypothesis to test.

8. The AGE tool used in family medicine is acceptable and feasible for patients and family practitioners

#### Hypothesis 8.1

At least 50% of physicians in the intervention arm used the BAT at least once

## Hypothesis 8.2

At least 50% of physicians in the intervention arm used the BAT at least once for all their patients included in the study

## Hypothesis 8.3

At least 50% of the patients included in the intervention arm had a BAT result







| SOP Plan d'analyse statistique | | |
|--------------------------------|---------------|----------------|
| SOP CRC-CHUV DM201 AN01 | | |
| Création : | Yolanda Mülle | r / 29.11.2018 |
| Révision : | | |
| Approbation: | IL. NS | |

#### Hypothesis 8.4

At least 50% of the patients who had a BAT once had a second BAT repeated after one year

#### Hypothesis 8.5

When using the BAT, physicians reported at least 50% of the items (4 out of 8 syndromes screened)

## Hypothesis 8.6

When using the BAT, physicians reported at least 87.5% of the items (7 out of 8 syndromes screened)

## Hypothesis 8.7

Agreement between BAT result and physician judgement was at least moderate (kappa >0.4) in suspecting geriatric syndromes

#### Hypothesis 8.8

A plan of care is completed in at least 50% of patients with a suspected geriatric syndrome

## Hypothesis 8.9

Adhesion to the recommendations of the plan of care is documented in at least 50% of patients with a suspected geriatric syndrome

#### Qualitative analysis

In addition, the following aspects will be evaluated in the qualitative analysis: acceptability and feasibility of the intervention, and of perceptions of autonomy in elderly patients and family physicians

## Safety:

9. The AGE tool administered in family medicine does not impact the quality of life, hospitalization and death rate of elderly patients.

#### Hypothesis 9.1:

The incidence rate of severe adverse events (SAE) (per person-year) in the intervention group does not exceed incidence rate in the control group (relative difference <10%)

#### Hypothesis 9.2:

The total WHOQOL-OLD score of patient in the intervention group is not inferior (difference<5 points on a transformed scale of 0 to 100) to the score of patients in the control group

## Hypothesis 9.3:

The admission rate (number of admission per person-year) in the intervention group does not exceed admission rate in the control group (relative difference <10%)

## Hypothesis 9.4:







| SOP Plan d'analys | e statistique | |
|-------------------------|-----------------------------|---------------|
| SOP CRC-CHUV DM201 AN01 | | |
| SOP AGE3 DM AN | 101 | Version : V01 |
| Création : | Yolanda Müller / 29.11.2018 | |
| Révision : | : | |
| Approbation: | IL, NS | |

The institutionalization rate (number of institutionalization per person-year) in the intervention group does not exceed institutionalization rate in the control group (relative difference <10%)

#### Hypothesis 9.5:

The death rate (number of deaths per person-year) in the intervention group does not exceed death rate in the control group (relative difference <10%)

## Economic analysis

#### Hypothesis 10.1

Use of the AGE tool increases in ambulatory costs (number of consultations, referrals, investigations)

## Hypothesis 10.2

Use of the AGE tool decreases medication costs

#### Hypothesis 10.3

Use of the AGE tool decreases the number of hospitalization, institutionalization, and use of home-based care

# 3. MODIFICATIONS OF STUDY OBJECTIVES DURING THE STUDY

Protocol amendment 04/09/2017, approved by CER-VD on 27.09.2017:

Preliminary analysis of baseline data of the first 247 patients showed that the majority of patients had a baseline IADL score of 8. Therefore, initial assumption of a mean score of 5 and use of a Poisson model were not appropriate anymore. We reformulated our hypothesis to show a difference in the proportion of patients not independent on IADL, i.e. patients that score less than 8 IADL[1]. Also, we refined the intraclass correlation estimation for the sample size calculation, because by contrast with our previous AGE1 and AGE2 study, IADL are assessed by a single rater in AGE3. However, the effect of the intervention itself might differ by FP, causing some degree of intracluster correlation after 2 years in the intervention arm.

However, after realizing that many men start below 8 not because of a loss of independence, but because they never performed some activities done by their spouse, we further reformulated our hypothesis to show a difference in "incident disability", i.e. patients that lose at least one IADL between baseline and after 2 years [1].

## 4. STUDY DESIGN

Controlled, open label, cluster randomized superiority trial. The unit of randomization is a family practitioner (FP). FP are recruited in french-speaking Switzerland and randomly allocated (1:1 ratio) to one of the two parallel arms (AGE or usual care). A total of 46 FP's will be recruited by arm. Ten







| SOP Plan d'ana | ılyse statistiqu | е |
|----------------|------------------|---------------------|
| SOP CRC-CI | HUV DM201 | 1 AN01 |
| Création : | Yolanda M | füller / 29.11.2018 |
| Révision : | | |
| Approbation: | IL, NS | |

patients aged 75 years and over will be recruited per FP. Therefore in total 46 FP's and 460 patients will be involved (see sample size estimate below). The follow-up of patients will be for 2 years per patient.

## Efficacy:

The AGE tool used in family medicine reduces the functional decline of elderly patients.
 Outcome: Activities of daily living (ADL) score and instrumental ADL (IADL) score

Source: Phone interview

Recoding: Category of patients with at least one loss of IADL, respectively ADL and IADL + ADL, between baseline and 2 years.

2. The AGE tool used in family medicine improves the quality of life of elderly patients. Outcome: Health related quality of life (WHOQOL-OLD) score

Six facets: 1) Sensory abilities, 2) Autonomy, 3) Past, present and future activities, 4) Social participation, 5) Death and dying and 6) Intimacy

Source: Phone interview

Recoding: according to WHO Manual (The WHOQOL-OLD module – manual, WHO European office, May 2006):

- Recoding of negatively worded items
- Summing items belonging to a facet (raw facet score; range 4 to 20)
- Standardising mean facet score (raw facet score divided by number of items, any decimal value between 1 and 5)
- Transferring to raw score to a transformed scale score between 0 and 100
- Similarly, adding the facet scores to constitute a total raw score, a total standardized mean score and a total transformed (0 to 100) score
- 3. The AGE tool used in family medicine reduces the incidence of hospital admissions Outcome: Incidence of hospital admissions (number of admission per person-year of follow-up) Source: FP medical record

Recoding: Exclusion of hospital admissions <24 hours (corresponding to ambulatory visits but reported by mistake in this section)

4. The AGE tool used in family medicine reduces the incidence of institutionalizations
Outcome: Incidence of institutionalization (number of institutionalization per person-year of follow-up)

Source: FP medical record

Recoding: none







| SOP Plan d'analys | e statistique | |
|------------------------------|---------------|----------------|
| SOP CRC-CHUV DM201 AN01 | | |
| SOP AGE3 DM AN01 Version : \ | | Version : V01 |
| Création : | Yolanda Mülle | r / 29.11.2018 |
| Révision : | | |
| Approbation: | IL, NS | |

5. The AGE tool used in family medicine reduces the incidence of emergency visits Outcome: Incidence of emergency visits (number of emergency visits per person-year of follow-up)

Source: FP medical record

Recoding: none

6. The AGE tool used in family medicine impacts on the number of FP outpatient visits Outcome: Incidence of outpatient visits (number of outpatient visits per person-year of follow-up) Source: FP medical record

Recoding: none

7. The AGE tool used in family medicine improves the processes of care (diagnoses and management) of elderly patients

#### Outcome:

- Number of geriatric syndromes identified, respectively confirmed, in intervention arm
- Number of new chronic conditions diagnosed after baseline, in particular:
  - o Rectal incontinence D17
  - New eye condition (entire F group, F83 (retinopathy), F84 (macular degeneration), F94 (blindness))
  - New ear condition (entire H group, H02 (hearing problem) H86 (deafness))
  - New transitory ischemic incident (H89), cerebrovascular event (H90), cerebrovascular disease (K91)
  - New osteoporosis (L95)
  - New urinary incontinence (U04)
  - o New dementia (P70), memory disorder (P20), depression (P76)
  - o New fracture (L72 to L76)
  - Source: Process questionnaire, data from medical records
- Comparison of a selected number of managements strategies between intervention and control arm
  - Hip replacement (medical record)
  - Knee replacement (medical record)
  - o Cataract intervention (medical record)
- Comparison of patient follow-up
  - Number of consultations
  - o Number of contact with family / helpers, physically or by phone
  - o Number of contact with home-based care
  - o Number of specialist referrals: ophthalmologist, gynaecologist, urologist, neurologist, geriatrician, rheumatologist, orthopedist, ENT, dentist, memory clinic, other.
  - Number of phone contact with geriatrician
  - Number of weight assessments
  - Number of height assessment
  - Clinical examination: neurological, osteoarticular, digestive, urogenital or anal, mouth, vision
  - Evaluation of alcohol consumption, nutrition (food intake), physical exercise
  - Score use: MMSE, Moca, GDS, IADL, other
  - Prescription of home-based care, physiotherapy, ergotherapy, pelvic physiotherapy,







| SOP Plan d'analys | e statistique | |
|-------------------------|---------------|-----------------|
| SOP CRC-CHUV DM201 AN01 | | |
| SOP AGE3 DM AN | N01 | Version : V01 |
| Création : Yolanda M | | er / 29.11.2018 |
| Révision : | | |
| Approbation: | II NS | |

urinary protection, physical exercise, nutrition supplements

- Comparison of investigations
  - Blood count, HbA1c, creatinine clearance, liver function tests, gammaGT, Na, K, Ca, vitamin B12, Folic acid, urinary stick, thyroid function, cerebral RMN, osteodensitometry
- Comparison of medication
  - o Number of patients on Calcium and/or vitamin D (A12AX00)
  - o Number of patients with biphosphonates
  - Number of patients on anticholinergic
  - Number of patients with antidepressant
  - Number of patients with precognitive medication
- Deprescription
  - Number of oral+ parenteral medication
  - Number of potentially inappropriate prescriptions (PIMs) according to 2015 Beers criteria
  - Specific PIMs (ATC code):
    - Benzodiazepines and other psychotropic medications (N05 N06)
    - Statins (C10A)
    - Drugs at risk orthostatic hypotension: peripheral and central alpha-1 blockers (C02CA)
    - Hypoglycaemic drugs (chlorpropamide A10BB02, glyburide A10BB01, insulin A10A)
- 8. The AGE tool used in family medicine is acceptable and feasible for patients and family practitioners

#### Outcome:

- Proportion of physicians in the intervention arm using the BAT at least once
- Proportion of physicians in the intervention arm using the BAT at least once for all their patients included in the study
- Proportion of physicians in the intervention arm using the BAT a second time, after using it the first time
- Proportion of use of the different items contained in the BAT
- Proportion of adhesion the different items contained in the plan of care, separated into investigatins and attitudes
- By section: proportion of FPs adhering to at least half of the recommended investigations, respectively attitudes
- Agreement between assessment by the BAT and by FP
- Qualitative analysis of acceptability and feasibility of the intervention, and of perceptions of autonomy in elderly patients and family physicians

#### Safety:

- 9. The AGE tool administered in family medicine does not impact the quality of life, hospitalization and death rate of elderly patients.
  - Outcome:

     Annual incidence of SAE between intervention and control arm (nb of events per person-year)
    - Recoding: SAE reviewed by study coordinator to check if really fitting SAE definition







| SOP Plan d'analyse statistique | | |
|---|---|---|
| SOP CRC-CHU | SOP CRC-CHUV DM201 AN01 | |
| Création : | Yolanda Mülle | r / 29.11.2018 |
| Révision : | | |
| Approbation: | IL, NS | |

- Annual incidence of admissions between intervention and control arm (nb of events per personvear)
- Annual mortality rate between intervention and control arm (nb of deaths per person-year)
- WHOQOL-OLD score between intervention and control arm

## Economic analysis

Outcome: incremental cost-effectiveness ratio par preserved ADL

#### Hypothesis 10.1

Use of the AGE tool increases in ambulatory costs

#### Outcomes:

- o Billing data of GPs for patients included in the study
- Number of consultations,
- o Number of referrals,
- Number of investigations

#### Hypothesis 10.2

Use of the AGE tool decreases medication costs

#### Outcomes:

- Prescription data by ATC-code
- Estimated cost difference between arms for medications with at least 5% difference in prescription by arm.

#### Hypothesis 10.3

Use of the AGE tool decreases the number of hospitalization, institutionalization, and use of home-based care

## Outcomes:

- o Number of hospitalizations
- Number of institutionalization
- Time to institutionalization
- Use of home-based care (use / no use and frequency of use)

# 5. POPULATION - SAMPLING

#### Sampling

The study will be conducted in primary care practices located in the canton of Vaud. Because target of FP recruitment proved difficult to achieve in only one canton, the study was extended to FPs working in other french-speaking cantons of Switzerland (Valais, Neuchâtel and Fribourg) in January 2017. The study is will be proposed to any patients aged 75 years or older being followed-up in a FP practice



consulting during the recruitment period. Before starting enrolment, FP decide whether they prefer to propose the study consecutively to all eligible patients until 12 are enrolled, or whether they prefer to propose the study to only one patient per consultation day, selected randomly. Random selection is done by tossing a coin (if two patients) or drawing a number from a bag containing numbered chips corresponding to the numbers of eligible patients.

Details about recruitment procedure and eligibility criteria can be found in the study protocol.

## Sample size calculation

In order to estimate the sample size needed for our purposes, we assumed that 10% of patients would lose independence in at least one activities (IADL) in the intervention group, compared with 25% in the control group. This is in line with what was observed in other similar interventional studies[2].

A mixed effect logistic model was adopted in order to describe data, with a doctor-related random effect. With these parameters, cluster data were generated with n FP's per group and m patients per FP (n = 5,10,...,55,60; m = 5,10,...,25,30). For each combination of n and m, 10'000 datasets were generated and the power was empirically calculated as the percentage of datasets on which a significant  $(\alpha=0.05)$ difference between the two arms was obtained via the logistic mixed effect model, for different levels of ICC. Results are shown in Figure 1. In the absence of available data of intracluster coefficient (ICC) for such a type of interventions, and with an ICC of 0 at baseline, we expect only a cluster effect in half of the participants after 2 years (intervention arm), which we postulated to be 0.10 considering the standardized nature of the intervention.



Figure 1. Simulation for sample size calculation

Version: V01







| SOP Plan d'analyse statistique | | |
|---|---|---|
| SOP CRC-CHU | SOP CRC-CHUV DM201 AN01 | |
| Création : | Yolanda Mülle | r / 29.11.2018 |
| Révision : | | |
| Approbation: | IL, NS | |

This approach allows choosing the best cluster combination that includes also feasibility considerations. For example to achieve a power of 90%, 8 patients per FP are sufficient if we have 20 FP's per arm, based on an ICC is 0.10. Taking into account the loss to follow-up estimated at 15%, we increased the number of patients per FP to 8/(1-0.15)=10, corresponding to a total of **40 FP's and 400 patients.** 

Sample size calculation was based on IADL because of the larger variance observed in this variable with respect to ADL on AGE 1 data. It represents therefore the "worst case scenario".

#### Qualitative sub-study

The study population for the qualitative evaluation is a subset of the AGE3 trial study population. We aim to recruit about 20 patients and 6 to 8 physicians, before reaching data saturation.

The sample size for patients has been estimated in order to cover the main patient constellations in terms of age, gender, support by home care, level of profession, and geography (rural/semi-urban/urban residence).

For physicians, we aim for a balanced age and sex distribution. In addition, we will consider group versus single practice and canton (Vaud versus other), as well as their practice location (rural/semi-urban/urban).

## Randomisation, arm allocation and blinding

#### Randomisation

The randomisation unit will be the family practitioner, allocated on a 1:1 ratio to the intervention or usual care group. Randomisation will take place during training sessions organised during half a day for FPs participating in the study.

Participating FPs will be given a unique ID at the time of the previsit by the study staff. An independent statistician generated a randomisation list based on uneven block size. He will then prepare sealed opaque envelopes containing the allocation arm, with a printed number (identification number, ID) on the outside. When attending the training session, the FP opened the envelope corresponding to his unique ID. The allocation lists (containing the identification number and allocation after each randomisation session) was kept in sealed envelopes by the PI.

#### Blinding procedures

FPs and study participants will be unblinded to their allocation. The study staff (medical assistant) performing the main outcome measures (phone interviews) is blinded to the allocation. The study coordinator in charge of study and data monitoring also is also blinded to the allocation. The study assistant that conducts the annual visits to the family practice is not blinded to the allocation. Data related to the BAT specifically will be monitored by the unblinded study assistant and an external statistician. The study statistician in charge of the interim and final analysis will be blinded to the allocation.

#### Allocation masking

Allocation will be recorded into the eCRF because this information is necessary to determine which forms the FP has to complete, but it will not be visible to users (study staff). The forms recording information on the AGE tool will not be accessible to users apart from FP and study assistant conducting annual visits. Data monitoring of AGE-specific sections will be performed on unlinked datatables, after recoding of the identifier by an external datamanager so that it cannot be linked to patient or FP. Queries will be transmitted back to the FP through this data manager.

Details about procedures to minimize risk of bias can be found in the study protocol.

| Policlinique<br>Médicale<br>Universitaire |
|-------------------------------------------|
|-------------------------------------------|





| SOP Plan d'analyse statistique | | |
|--------------------------------|--------|-----------------|
| SOP CRC-CHUV DM201 AN01 | | |
| SOP AGE3 DM AN01 Version : V0 | | |
| Création : Yolanda M | | er / 29.11.2018 |
| Révision : | | |
| Approbation: | IL. NS | |

## 6. GLOSSARY OF STUDY VARIABLES

#### Main outcomes:

- Activities of daily living (ADL) score and instrumental ADL (IADL) score[3, 4] The use of (instrumental) "activities of daily living" scales (IADL and ADL) is the simplest and most reliable way to assess functional decline. According to previous studies using this outcome in similar populations, one point (= one activity) lost avoided out of 8 activities (for IADL) over 1 year can be considered as a significant and meaningful improvement.[2, 5] These two instruments have been used in numerous studies, are sensitive to change and foremost can be reliably administered by phone[6, 7]. Although very frequently used, psychometric properties of this scale can be questioned, in particular because of a marked ceiling effect [8]. Also, many items of the classic ADL scales are gender-specific, and reduced scores can be more related to traditional roles in society more than actual disability.
- Health related quality of life (WHOQOL-OLD) score [9, 10]
- This broadly validated instrument is composed of six facets: 1) Sensory abilities, 2) Autonomy, 3) Past, present and future activities, 4) Social participation, 5) Death and dying and 6) Intimacy. [10] Like with ADL and IADL, this questionnaire can be administered by phone. Pre-post intervention studies testing the effect of hearing aids and cardiac surgery among elderly people have reported improvements between 2 and 8 points/100[11-14]. Comparisons of mean scores were usually based on paired t-tests, sometimes also used adjusted linear models. One study has compared the proportion of patients with improved / no change / worsened WHOWOL-OLD score[11]. We found no population-based data reporting longitudinal evolution of WHOQOL-OLD score in the absence of intervention.

| Variable<br>name | Data table | Variable<br>type :<br>Categoric,<br>ordinal,<br>quantitative | Modalities (coding) | Description | Recodin |
|---|---|---|---|---|---|
| tel | 5.Téléphone | Ordinal | 1 Vous utilisez le téléphone de votre propre initiative, cherchez les numéros, appelez, répondez, etc. 2 Vous n'appelez que quelques numéros bien connus 3 Vous répondez au téléphone, mais n'appelez pas 4 Vous n'utilisez pas le téléphone 9 Ne sait pas / ne veut pas répondre / non évaluable | IADL | 1/3=1 4=<br>9=. |







SOP Plan d'analyse statistique SOP CRC-CHUV DM201 AN01

Programme AGE Centre de recherche et développement
PMU | Policlinique médicale universitaire
Rue du Bugnon 44 | BU44 04-2316
1011 Lausanne | Suisse
Tél 021 314 32 94 ou 079 556 11 48

Version: V01 SOP AGE3 DM AN01 Yolanda Müller / 29.11.2018 Création: Révision: IL, NS Approbation:

| comm | 5.Téléphone | Ordinal | 1 Vous vous occupez de tous les achats et commissions, indépendamment 2 Vous vous occupez uniquement de petits achats 3 Vous avez besoin d'être accompagné(e) pour chaque commission 4 Vous êtes complètement incapable de faire vos commissions 9 Ne sait pas / ne veut pas répondre / | IADL | 1=1 2/4=<br>9=. |
|---|---|---|---|---|---|
| repas | 5.Téléphone | Ordinal | non évaluable 1 Vous planifiez, préparez et servez des repas adéquats, de façon indépendante 2 Vous préparez des repas adéquats, pour autant que la matière première soit fournie 3 Vous réchauffez des repas ou préparez des repas MAIS ne maintenez pas une diète adéquate 4 Vous avez besoin d'avoir des repas préparés et servis 9 Ne sait pas / ne veut pas répondre / non évaluable | IADL | 1=1 2/4=<br>9=. |
| menage | 5.Téléphone | Ordinal | 1 Vous vous occupez du ménage seul(e) ou avec de l'assistance occasionnelle (p.ex. travaux de réparation lourds) 2 Vous vous occupez seulement de tâches ménagères légères comme laver la vaisselle ou faire le lit 3 Vous vous occupez seulement de tâches ménagères légères MAIS êtes incapables de maintenir un niveau de propreté adéquat 4 Vous nécessitez de l'assistance pour toutes les tâches ménagères, mais vous participez 5 Vous ne participez pas aux tâches ménagères 9 Ne sait pas / ne veut pas répondre / | IADL | 1/4=1 5=<br>9=. |
| lessive | 5.Téléphone | Ordinal | non évaluable 1 Vous faites toute votre lessive 2 Vous ne vous occupez que de « petite lessive » (p.ex. chaussettes, etc) 3 Toute la lessive doit être faite par d'autres personnes 9 Ne sait pas / ne veut pas répondre / non évaluable | IADL | 1/2=1 3=<br>9=. |



| transports | 5.Téléphone | Ordinal | 1 Vous voyagez indépendamment en utilisant les transports publics ou votre | IADL | 1/3=1<br>4/5=0 9= |
|---|---|---|---|---|---|
| | | | propre voiture 2 Vous voyagez indépendamment en taxi MAIS n'utilisez pas d'autres transports publics 3 Vous voyagez en utilisant les transports publics MAIS uniquement lorsqu'accompagné-e 4 Vous voyagez uniquement en taxi ou | | |
| | | | automobile et avec accompagnement<br>5 Vous ne voyagez pas du tout<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | | |
| medic | 5.Téléphone | Ordinal | 1 Vous êtes entièrement responsable de prendre vos médicaments à dose correcte et horaire prescrit 2 Vous êtes responsable de prendre vos médicaments s'ils sont préparés à l'avance en doses séparées | IADL | 1=1 2/3=<br>9=. |
| | | | <ul><li>3 Vous êtes incapable de prendre seul-e<br/>vos médicaments</li><li>9 Ne sait pas / ne veut pas répondre /<br/>non évaluable</li></ul> | | |
| finances | 5.Téléphone | Ordinal | 1 Vous vous occupez de vos paiements et finances indépendamment (vous payez le loyer, faites vos paiements, etc.) 2 Vous vous occupez des paiements quotidiens, MAIS nécessitez de l'aide pour maintenir les autres 3 Vous êtes incapable de vous occuper des paiements 9 Ne sait pas / ne veut pas répondre / non évaluable | IADL | 1/2=1 3=<br>9=. |
| hygiene | 5.Téléphone | Ordinal | 1 Vous ne recevez aucune assistance 2 Vous recevez de l'assistance pour laver une partie du corps (dos ou jambes) 3 Vous recevez de l'assistance pour laver plus qu'une partie du corps 9 Ne sait pas / ne veut pas répondre / | bADL | 1/2=1 3=<br>9=. |
| habil | 5.Téléphone | Ordinal | non évaluable 1 Vous prenez vos habits de l'armoire et des tiroirs et vous vous habillez sans assistance 2 Vous prenez vos habits de l'armoire et des tiroirs et vous vous habillez sans assistance, à l'exception des chaussures 3 Vous recevez de l'assistance pour prendre vos habits, ou pour vous habiller, ou vous ne vous habillez pas vous-mêmes | bADL | 1/2=1 3=<br>9=. |



Programme AGE





SOP Plan d'analyse statistique

# SOP CRC-CHUV DM201 AN01

SOP AGE3 DM AN01

Version : V01

Centre de recherche et développement
PMU | Policlinique médicale universitaire

Rue du Bugnon 44 | BU44 04-2316 1011 Lausanne | Suisse Tél 021 314 32 94 ou 079 556 11 48 Révision :

Yolanda Müller / 29.11.2018

Création : Révision :

Approbation: IL, NS

9 Ne sait pas / ne veut pas répondre / non évaluable

| toilet | 5.Téléphone | Ordinal | 1 Vous allez aux toilettes, vous vous nettoyez et vous vous rhabillez sans | bADL | 1=1 2/3=<br>9=. |
|---|---|---|---|---|---|
| | | | assistance 2 Vous recevez de l'assistance pour aller aux toilettes ou pour vous nettoyer après ou pour vous rhabiller ou pour l'utilisation du vase, de l'urinal ou de la chaise percée 3 Vous ne pouvez pas utiliser les toilettes 9 Ne sait pas / ne veut pas répondre / non évaluable | | |
| transfert | 5.Téléphone | Ordinal | 1 Vous sortez, entrez dans le lit ou d'une chaise sans assistance (peut utiliser une canne ou un déambulateur) 2 Vous sortez et entrez dans le lit ou d'une chaise avec assistance seulement 3 Vous ne sortez pas du lit 9 Ne sait pas / ne veut pas répondre / non évaluable | bADL | 1=1 2/3=<br>9=. |
| continence | 5.Téléphone | Ordinal | 1 Vous contrôlez urine et selles totalement de vous-même 2 Vous avez des « accidents » occasionnels 3 Vous nécessitez une supervision pour rester propre ou vous nécessitez un cathéter, ou vous êtes incontinent 9 Ne sait pas / ne veut pas répondre / non évaluable | bADL | 1=1 2/3=<br>9=. |
| aliment | 5.Téléphone | Ordinal | 1 Vous vous nourrissez sans assistance 2 Vous vous nourrissez seul mais nécessitez de l'assistance pour couper la viande ou beurrer le pain 3 Vous recevez de l'assistance pour vous nourrir ou vous êtes nourri partiellement ou complètement par sonde ou en parentéral (intraveineux) 9 Ne sait pas / ne veut pas répondre / non évaluable | bADL | 1/2=1 3=<br>9=. |







SOP Plan d'analyse statistique

SOP CRC-CHUV DM201 AN01 SOP AGE3 DM AN01

Version: V01

Programme AGE
Centre de recherche et développement
PMU | Policlinique médicale universitaire
Rue du Bugnon 44 | BU44 04-2316
1011 Lausanne | Suisse
Tél 021 314 32 94 ou 079 556 11 48

Création: Révision:

Yolanda Müller / 29.11.2018

IL, NS Approbation:

| f25_1 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu,<br>3 Modérément, 4 Beaucoup<br>5 Enormément<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=.<br>4=; |
|---|---|---|---|---|---|
| f25_3 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu,<br>3 Modérément, 4 Beaucoup<br>5 Enormément<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=.<br>4=; |
| f26_1 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu<br>3 Modérément, 4 Beaucoup<br>5 Extrêmement<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=. |
| f26_2 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu<br>3 Modérément, 4 Beaucoup<br>5 Extrêmement<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=. |
| f26_4 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu<br>3 Modérément, 4 Beaucoup<br>5 Extrêmement<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=. |
| f29_2 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu<br>3 Modérément, 4 Beaucoup<br>5 Extrêmement<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=.<br>4=; |
| f29_3 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu<br>3 Modérément, 4 Beaucoup<br>5 Extrêmement<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=.<br>4=; |
| f29_4 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu<br>3 Modérément, 4 Beaucoup<br>5 Extrêmement<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=.<br>4=: |



| SOP Plan d'analyse statistique | | |
|---|---|---|
| SOP CRC-CHL | SOP CRC-CHUV DM201 AN01 | |
| Création : Yolanda Mülle | | er / 29.11.2018 |
| Révision : | : | |
| Approbation: | II NS | |

| f29_5 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu<br>3 Modérément, 4 Beaucoup<br>5 Extrêmement<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=.<br>4=; |
|---|---|---|---|---|---|
| f25_4 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu<br>3 Modérément, 4 Beaucoup<br>5 Entièrement<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=.<br>4=; |
| f26_3 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu<br>3 Modérément, 4 Beaucoup<br>5 Entièrement<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=. |
| f27_3 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu<br>3 Modérément, 4 Beaucoup<br>5 Entièrement<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=. |
| f27_4 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu<br>3 Modérément, 4 Beaucoup<br>5 Entièrement<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=. |
| f28_4 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu<br>3 Modérément, 4 Beaucoup<br>5 Entièrement<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | ー <u></u><br>f28<br>f28 |
| f27_5 | 5.Téléphone | Ordinal | 1 Très insatisfait-e, 2 Insatisfait-e<br>3 Ni satisfait-e, ni insatisfait-e<br>4 Satisfait-e, 5 Très satisfait-e<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=. |
| f28_1 | 5.Téléphone | Ordinal | 1 Très insatisfait-e, 2 Insatisfait-e<br>3 Ni satisfait-e, ni insatisfait-e<br>4 Satisfait-e, 5 Très satisfait-e<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=. |







SOP Plan d'analyse statistique

SOP CRC-CHUV DM201 AN01

IL, NS

SOP AGE3 DM AN01

Version: V01

Yolanda Müller / 29.11.2018

Programme AGE
Centre de recherche et développement
PMU | Policlinique médicale universitaire
Rue du Bugnon 44 | BU44 04-2316
1011 Lausanne | Suisse
Tél 021 314 32 94 ou 079 556 11 48

Approbation:

Création: Révision:

MILOCOL OLD

| f28_2 | 5.Téléphone | Ordinal | 1 Très insatisfait-e, 2 Insatisfait-e<br>3 Ni satisfait-e, ni insatisfait-e<br>4 Satisfait-e, 5 Très satisfait-e<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=. |
|---|---|---|---|---|---|
| f28.7 | 5.Téléphone | Ordinal | 1 Très insatisfait-e, 2 Insatisfait-e<br>3 Ni satisfait-e, ni insatisfait-e<br>4 Satisfait-e, 5 Très satisfait-e<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=. |
| f27.1 | 5.Téléphone | Ordinal | 1 Très malheureux/se, 2 Malheureux/se 3 Ni heureux/se, ni malheureux/se 4 Heureux/se, 5 Très heureux/se 9 Ne sait pas / ne veut pas répondre / non évaluable | WHOQOL-OLD | 9=. |
| f25.2 | 5.Téléphone | Ordinal | 1 Très mauvais, 2 Mauvais<br>3 Ni bon, ni mauvais, 4 Bon<br>5 Très bon<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=. |
| f30.2 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu,<br>3 Modérément, 4 Beaucoup<br>5 Enormément<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=. |
| f30.3 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu<br>3 Modérément, 4 Beaucoup<br>5 Extrêmement<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=. |
| f30.4 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu<br>3 Modérément, 4 Beaucoup<br>5 Entièrement<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=. |
| f30.7 | 5.Téléphone | Ordinal | 1 Pas du tout, 2 Un peu<br>3 Modérément, 4 Beaucoup<br>5 Entièrement<br>9 Ne sait pas / ne veut pas répondre /<br>non évaluable | WHOQOL-OLD | 9=. |







| SOP Plan d'analyse statistique | | |
|--------------------------------|---------------|-----------------|
| SOP CRC-CHUV DM201 AN01 | | |
| SOP AGE3 DM AN | V01 | Version : V01 |
| Création : | Yolanda Mülle | er / 29.11.2018 |
| Révision : | | |
| Approbation: | IL. NS | |

Composite variables:

Email Dmir ano@bosavid ah

| Composite va | riables: | | |
|---|---|---|---|
| Variable name | Data table | Variable type: Categoric, ordinal, quantitative | Modalities (coding) |
| avqi | 5.Téléphone | Ordinal | Avqitel +avqicomm +avqirepas +avqimenage +avqilessive +avqitranspo<br>+avqimedic +avqifinances |
| avqb | 5.Téléphone | Ordinal | avqbhygiene +avqbhabil+avqbtoilet +avqbtransfert+avqbcontinence+av |
| avqtot | 5.Téléphone | Ordinal | avqi+avqb |
| OLD_SAB_s | 5.Téléphone | Ordinal | f25_1_rec+ f25_3_rec+ f25_4_rec+ f25_2 |
| OLD_AUT_s | 5.Téléphone | Ordinal | f26_1 +f26_2 +f26_4 +f26_3 |
| OLD_PPF_s | 5.Téléphone | Ordinal | f27_3 +f27_4 +f27_5 +f27_1 |
| OLD_SOP_s | 5.Téléphone | Ordinal | f28_4+ f28_1 +f28_2 +f28_7 |
| OLD_DAD_s | 5.Téléphone | Ordinal | f29_2_rec +f29_3_rec +f29_4_rec +f29_5_rec |
| OLD_INT_s | 5.Téléphone | Ordinal | f30_2 +f30_3 +f30_4 +f30_7 |
| OLD_*_m | 5.Téléphone | Quantitative | Mean scores (1 to 5) |
| OLD_*_t | 5.Téléphone | Quantitative | Standardized scales (0 to 100) = 100*(mean score – 1)/4 |
| OLD_total_s | 5.Téléphone | Ordinal | OLD_SAB_s+OLD_AUT_s+OLD_PPF_s+OLD_SOP_s+OLD_DAL_+ |
| OLD_total_n | 5.Téléphone | Ordinal | anycount(f25_1_rec f25_3_rec f25_4_rec f25_2 f26_1 f26_2 f26_4 f26_ f27_3 f27_4 f27_5 f27_1 f28_4 f28_1 f28_2 f28_7 f29_2_rec f29_4_rec f29_5_rec /// f30_2 f30_3 f30_4 f30_7), values(1/5) |
| OLD_total_m | 5.Téléphone | Quantitative | OLD_total_s/OLD_total_n |
| OLD_total_t | 5.Téléphone | Quantitative | Standardized scales (0 to 100) = 100*(mean score – 1)/4 |

## Outcomes 3 to 6:

- Incidence of hospital admissions (number of admission per person-year of follow-up)
- Incidence of institutionalizations (number of institutionalizations per person-year of follow-up)
- Incidence of emergency visits (number of emergency visits per person-year of follow-up)
- Number of FP outpatient visits







SOP Plan d'analyse statistique

SOP CRC-CHUV DM201 AN01


Création : Yolanda Müller / 29.11.2018

Révision :

Approbation: IL, NS

Programme AGE
Centre de recherche et développement
PMU | Policlinique médicale universitaire
Rue du Bugnon 44 | BU44 04-2316
1011 Lausanne | Suisse
Tél 021 314 32 94 ou 079 556 11 48

6.Processus

| Email Day 200 | hanned ah | | Approbation: | IL, NS | |
|---|---|---|---|---|---|
| Variable<br>name | Data table | Variable<br>type :<br>Categoric,<br>ordinal,<br>quantitativ | | Description | Recodin |
| dateinc | 3.Inclusion | Date | | Date of inclusion | - |
| datefin | 8.FinSuivi | Date | | Date of end of follow-up | Actual da decision follow-up withdraw correspo datefin, i cas it is recoded. |
| Hospit | 6.Processus | Binary | 1 Oui, 0 Non,<br>9 Ne sait pas | Any admission | death be Recodec stohosp- (less tha |
| Institcourt | 6.Processus | Binary | 1 Oui, 0 Non,<br>9 Ne sait pas | Any short institutional stay | |
| institlong | 6.Processus | Binary | 1 Oui, 0 Non,<br>9 Ne sait pas | Any long institutional stay | |
| cslt | 6.Processus | Binary | 1 Oui, 0 Non,<br>9 Ne sait pas | Any emergency consultation | |
| Composite | variables: | | | | |
| Variable name | Data table | Variable<br>type :<br>Categoric,<br>ordinal,<br>quantitative | Modalities (coding) | | Description |
| Futime | : | Quantitative | Datefin-dateinc | | Duration o<br>follow-up in<br>the study |
| Nhosp | e_6_proc_hosp<br>bloc within<br>6.Processus | Quantitative | Sum of number of hospitalis | sation | |
| ninstit | e_6_proc_instit | Quantitative | Sum of number of short ins | titutional stays + institlong | |







SOP Plan d'analyse statistique

SOP CRC-CHUV DM201 AN01


Création : Yolanda Müller / 29.11.2018

Programme AGE
Centre de recherche et développement
PMU | Policlinique médicale universitaire
Rue du Bugnon 44 | BU44 04-2316
1011 Lausanne | Suisse
Tél 021 314 32 94 ou 079 556 11 48

Création : Yolanda Müller / 29.11.2018

Révision : IL, NS

| ncons | e_6_proc_cons | Quantitative | Sum of FP consultations |
|-------|---------------|--------------|-------------------------|
| | bloc within | | |
| | 6.Processus | | |

## **Process of care outcomes**

| Variable name | Data table | Variable<br>type :<br>Categoric,<br>ordinal,<br>quantitative | Modalities<br>(coding) | Description | Red |
|---|---|---|---|---|---|
| dateinc | 4.egb | Date | | Number of geriatric syndromes identified, respectively confirmed, in intervention arm | |
| datefin | 8.FinSuivi | Date | | Date of end of follow-up | Act |
| datemi | o.i iliodivi | Date | | bate of one of follow up | dec<br>follo |
| | | | | | (co<br>with<br>not |
| | | | | | to d<br>whi<br>ma |
| | | | | | rec<br>=da<br>of dat |
| Hospit | 6.Processus | Binary | 1 Oui, 0 Non,<br>9 Ne sait pas | Any admission | sto<br>sta<br>tha |
| Institcourt | 6.Processus | Binary | 1 Oui, 0 Non,<br>9 Ne sait pas | Any short institutional stay | |
| institlong | 6.Processus | Binary | 1 Oui, 0 Non,<br>9 Ne sait pas | Any long institutional stay | |
| csit | 6.Processus | Binary | 1 Oui, 0 Non,<br>9 Ne sait pas | Any emergency consultation | |
| Contpro | 6.Processus | Binary | 1 Oui, 0 Non,<br>9 Ne sait pas | Au cours de l'année écoulée, selon le dossier médical, le médecin a-t-il eu contact avec les proches, physiquement ou par téléphone? | |







SOP Plan d'analyse statistique

SOP CRC-CHUV DM201 AN01


Création : Yolanda Müller / 29.11.2018

Révision :

Approbation: IL, NS

Programme AGE
Centre de recherche et développement
PMU | Policlinique médicale universitaire
Rue du Bugnon 44 | BU44 04-2316
1011 Lausanne | Suisse
Tél 021 314 32 94 ou 079 556 11 48

| Contprophys | 6.Processus | Quantitative | AND | |
|---|---|---|---|---|
| | | | | Nombre d'entretiens face-à-face |
| contprotel | 6.Processus | Quantitative | | Nombre d'entretiens téléphoniques |
| Contems | 6.Processus | Quantitative | | Contact with home-based care |
| ncontcms | 6.Processus | Quantitative | | Number of contact with home-based care (contcmsphys+contcmstel+contcmslet) |
| ophtalmo | 6.Processus | Binary | | |
| gyneco uro neuro geriatr rhumato ortho orl dentiste memoir specaut | | | | Number of specialist referrals: ophthalmologist, gynaecologist, urologist, neurologist, geriatrician, rheumatologist, orthopedist, ENT, dentist, memory clinic, other. |
| contgertel | 6.Processus | Quantitative | | Number of phone contact with geriatrician |
| exneuro<br>exos<br>exdig<br>exuro<br>exdent | 6.Processus | Binary | 1 Oui, 0 Non,<br>9 Ne sait pas | Clinical examination: neurological, osteoarticular, digestive, urogenital or anal, mouth, vision |
| exvis evalof evalalim evalexe | 6.Processus | Binary | 1 Oui, 0 Non,<br>9 Ne sait pas | Evaluation of alcohol consumption,<br>nutrition (food intake), physical<br>exercise |
| scmmse<br>scmoka<br>scgds<br>scavqi<br>scaut | 6.Processus | Binary | 1 Oui, 0 Non,<br>9 Ne sait pas | Score use: MMSE, Moca, GDS, IADL, other |
| ordcms ordergo ordphys ordspec ordurin ordex ordprot ordaut* | 6.Processus | Binary | 1 Oui, 0 Non,<br>9 Ne sait pas | Prescription of home-based care, physiotherapy, ergotherapy, pelvic physiotherapy, urinary protection, physical exercise, nutrition supplements |
| fs<br>hba1c<br>clair | 6.Processus | Binary | 1 Oui, 0 Non,<br>9 Ne sait pas | Comparison of investigations o Blood count, HbA1c, creatinine clearance, |





SOP Plan d'analyse statistique SOP CRC-CHUV DM201 AN01 Version: V01 SOP AGE3 DM AN01 Yolanda Müller / 29.11.2018 Création: Révision: IL, NS

Programme AGE Centre de recherche et développement PMU | Policlinique médicale universitaire Rue du Bugnon 44 | BU44 04-2316 1011 Lausanne | Suisse Tél 021 314 32 94 ou 079 556 11 48

liver function tests, asat gammaGT, Na, K, Ca, ggt vitamin B12, Folic nak acid, urinary stick, ca thyroid function, b12 cerebral RMN, folate osteodensitometry stix thyr irm densito

Approbation:

| Variable name | Data table | Variable type | Modalities (coding) | Description |
|---|---|---|---|---|
| | | Categoric,<br>ordinal,<br>quantitative | | |
| Nsynd | 4.egb | Discrete | urin dep cog vis aud chut osteo denut if (tot'x'==1 tot'x'ver==1) +1 if ((chute==1 marche==1)) & totchut!=1 & totchutver!=1 | Number of geri<br>syndromes ider<br>intervention arr<br>to BAT (tot) or<br>FP (ver) |
| Nsyndconf | 4.egb /<br>6.Processus | Discrete | Sum of: - New ccu04 diagnosis (urinary incontinence) - Confirmed depression depconf or new ccp76 - Confirmed cognitive disorder cogconf or new ccp70 or ccp20 - New eye condition (entire F group, F83 | Number of new<br>geriatric syndro<br>intervention arr<br>control arm but<br>EGB var) |
| | | | <ul> <li>retinopathy), F84 (macular degeneration), F94 (blindness))</li> <li>New ear condition (entire H group, H02 (hearing problem) H86 (deafness))</li> <li>Chute OR marche</li> <li>Fracture OR new osteoporosis (ccl95) OR new fracture L72 to L76</li> <li>Denutrition (T08 OR T91? Not optimal!)</li> </ul> | |
| Pthnew | 6.Processus | Binary | Pth (end) – pth (baseline) | Number of pati<br>new hip replace<br>baseline |
| Ptgnew | 6.Processus | Binary | Ptg (end) – ptg (baseline) | Number of pati<br>new knee repla<br>since baseline |
| Catanew | 6.Processus | Binary | Cataract (end) – cataract (baseline) | Number of pati<br>new hip replace<br>baseline |
| Npoids | e_6_proc_cons<br>6.Processus | Discrete | | Number of we assessments |
| nweight | e_6_proc_cons<br>6.Processus | Discrete | : | Number of he assessment |







SOP Plan d'analyse statistique

SOP CRC-CHUV DM201 AN01


Création : Yolanda Müller / 29.11.2018

Révision :

IL, NS

Programme AGE
Centre de recherche et développement
PMU | Policlinique médicale universitaire
Rue du Bugnon 44 | BU44 04-2316
1011 Lausanne | Suisse
Tél 021 314 32 94 ou 079 556 11 48

| nbmed | 12.Traitement | Discrete | | Number of or |
|---|---|---|---|---|
| | | | | parenteral me |
| nbcat | 12.Traitement | Categorical | 1 "0-4" 2 "5-9" 3 "10-14" 4 "15+" | Category of |
| | | | | polymedicatic<br>Number of pa |
| maxA12AX00 | 12.Traitement | Binary | | Calcium and/ |
| | | | | D Calcium and/ |
| | | | | Б |
| maxM05B | 12.Traitement | Binary | | Number of pa |
| Maxiviosb | 12. Haitement | Diricity | | bisphosphona |
| | | | | other drugs a |
| | | | | bone minerali |
| | | | | bone structure |
| ? | 12.Traitement | Binary | | Number of pa |
| | | | | anticholinergi- |
| maxN06A | 12.Traitement | Binary | | Number of pa |
| | | | | antidepressar |
| maxN06D | 12.Traitement | Binary | | Number of pa |
| Maxivood | 12. Haitement | Diricity | | precognitive r |
| npim | 12.Traitement | Discrete | Manual recoding from David | Number of pc |
| | 12.11. | | | inappropriate |
| | | | | prescriptions |
| | | | | according to 2 |
| | | | | criteria |
| maxN06A | 12.Traitement | Binary | | Number of pa |
| | | | | antidepressar |
| maxN05 | 12.Traitement | Binary | | Specific PIM: |
| maxN06 | 12. Hallomone | | | Benzodiazepi |
| | | | | other psychot |
| | | | | medications |
| maxC10A | 12.Traitement | Binary | | Specific PIM: |
| maxC02CA | 12.Traitement | Binary | | Specific PIM: |
| | | | | risk orthostati |
| | | | | hypotension: |
| | | | | and central al<br>blockers |
| | | | | Specific PIM: |
| maxA10BB01 | 12.Traitement | Binary | | Hypoglycaem |
| maxA10BB02 | | | | (chlorpropam |
| maxA10A | | | | A10BB02, gly |
| | | | | A10BB02, gry<br>A10BB01, ins |
| | 12.Traitement | Binary | | Specific PIM: |
| | ız. Hallement | Dirial y | | - |

Approbation:







SOP Plan d'analyse statistique

SOP CRC-CHUV DM201 AN01


Création : Yolanda Müller / 29.11.2018

Révision :

IL, NS

Programme AGE
Centre de recherche et développement
PMU | Policlinique médicale universitaire
Rue du Bugnon 44 | BU44 04-2316
1011 Lausanne | Suisse
Tél 021 314 32 94 ou 079 556 11 48

## Feasibility and acceptability outcomes

## Composite variables

| Description |
|---|
| Proportion of in the interverusing the BA once |
| egb not Proportion of inclusion in the intervusing the BA once for all the included in the |
| egb not Proportion of inclusion in the interverusing the BA time, after usifirst time |
| Proportion of<br>different items<br>contained in t |
| _ |

Approbation:







| SOP Plan d'analyse statistique | | |
|---|---|---|
| SOP CRC-CHUV DM201 AN01 | | |
| SOP AGE3 DM AN | NO1 | Version : V01 |
| Création : | Yolanda Müller / 29.11.2018 | |
| Révision : | | |
| Approbation: | IL, NS | |

| Not detailed | 4.EGB | this manufacture and a second discount of the second secon | Proportion of |
|---|---|---|---|
| not dotanoa | | | the different it |
| | | | contained in t |
| | | | care, separate |
| | | | investigations |
| | | | attitudes |
| Not detailed | 4.EGB | | By section: pr |
| | | | FPs adhering |
| | | | half of the |
| | | | recommende |
| | | | investigations |
| | | | respectively a |
| Tot*acc and | 4.EGB | | Agreement be |
| tot*ver | | | assessment t |
| | | | and by FP |

# Safety outcomes

Composite variables

| Variable name | Data table | Variable<br>type : | Modalities (coding) | Description |
|---|---|---|---|---|
| totSAE | 11.SAE / logSAE | Quantitative | Recoding: SAE reviewed by study coordinator to check if really fitting SAE definition | Annual incide between i and control a events per pe |
| Death | 11.SAE | Binary | 11.SAE:Categsae==1 OR 8.FinSuivi: motif==1 | Annual mor |
| | | | Manual recoding if death info but no record in SAE, and according to date of death | between i<br>and control a<br>deaths per pe |

# Economic analysis:

Variables included in "process of care", and billing data

| Variable name | Data table | Variable<br>type :<br>Categoric,<br>ordinal,<br>guantitative | Modalities (coding) | Description |
|---|---|---|---|---|
| totmontprest | 13.prestation | Quantitative | Sum of all montprest | Sum of all bille<br>between inclus<br>of follow-up |







| SOP Plan d'anal | yse statistiqu | e |
|-----------------|----------------|---------------------|
| SOP CRC-CH | IUV DM201 | AN01 |
| SOP AGE3 DM / | AN01 | Version : V01 |
| Création : | Yolanda M | lüller / 29.11.2018 |
| Révision : | : | |
| Approbation: | IL, NS | |

## 7. STATISTICAL ANALYSES

## 7.1 INTERMEDIATE ANALYSES

Analysis of baseline data will be conducted by the coPI once recruitment is complete. Mean and variance of IADL were assessed in slightly different patient populations than the AGE3 study population. If the analysis of baseline data shows important discrepancies compared to the assumptions made for the initial sample size calculation (baseline IADL, intra-class correlation), a new sample size estimation may be performed. If recruitment of additional FPs is needed to need sufficient power, this will be discussed with the steering committee and the protocol will be amended accordingly.

One interim analysis will be performed when at least 50% of patients have had their one year assessment. The interim analysis will be performed by the study statistician. If a difference on the main outcome (IADL) superior to the one expected after two years (difference in proportion having lost at least 1 IADL>15%) is observed between the two groups, the code will be broken and if it is shown that the difference is in favor of the intervention arm, the AGE tool will be offered to the patients of the usual care group. This decision will be made in collaboration with the steering committee. No futility rule is planned, as we acknowledge that the effect of the intervention may be somewhat delayed and therefore not necessarily apparent after one year only.

An annual safety analysis will be done by the study coordinator, comparing the incidence of hospital admissions and deaths between both groups. This will be included in the annual safety report submitted to the steering committee and the Ethics committee.

If there is a significant difference (p<0.05) between the two groups in terms of hospital admissions and deaths, the steering committee can decide to halt the study.

## 7.2 FINAL DATA ANALYSIS

## 7.2.1 Data management

#### **Dataset**

The AGE3 dataset consists of 685 variables for approximately 460 patients, organized in 13 study-specific forms.

#### **Forms**

- 0. Contact
- 1. Médecin
- Screening
- 3. Inclusion
- 4. EGB (Evaluation Gériatrique Brève)
- 5. Téléphone
- 6. Processus
- 7. Visites
- 8. FinSuivi







| SOP Plan d'analyse statistique | | |
|--------------------------------|--------|-----------------|
| SOP CRC-CHUV DM201 AN01 | | |
| Création : Yolanda Müll | | er / 29.11.2018 |
| Révision : | | |
| Approbation: | IL. NS | |

- 9. PlanSoins
- 11. SAE
- 12. Traitement
- 13. Prestations

Data are specified in an excel file describing each variable, variable label, type, value label, condition, limits and error messages.

Volume: Aug2017: 288 Ko for Raw data (zipped csv file), 1.4 Mo for .dta files.

Expected volume at the end of study: 1 Mo for raw data. Storage volume for incremental monthly extracts: about 1 Go

#### Qualitative evaluation

- Audio files and transcripts of patient observation, physician interviews and patient interviews
- MaxQDA files

#### Data collection:

The AGE3 database was designed using the secuTrial software, version 4.8.0.19. Data are stored in an Oracle database (v11), managed by the Informatic System Department of the CHUV, Lausanne.

#### Access:

The data manager has access to all study data (raw data extracts) and is in charge of preparing these extracts for data monitoring and analysis. In particular, he will remove contact details, recode age in years and remove date of birth, and unlink BAT and AGE related information from the unique identifier.

He has no role in data analysis per se.

The study statistician cannot enter or modify data but has access to all the study data, except contact details. BAT and AGE plan of care (which would reveal allocation) will only be linked to specific patients after completion of the ITT analysis.

## Electronic and central data validation

AGE3 data are collected via secuTrial.

Predefined checks incorporated in secuTrial are: concern mainly

- Respect of the time intervals between annual study visits.
- Height (>= 120 and <220 cm)

Secutrial software has an inbuilt data management tool allowing investigators to produce queries. Each form is revised by a member of the study staff. After solving of the pending queries, each form is locked, preventing further modification.

Completion status of each section was predefined during database development. The secuTrial system includes visual aid to inform of data entry completion.

Monthly exports of the data as .csv files are performed by the data manager and stored in her personal folder. Data are then transformed to respect anonymisation (excluding Contact information) and blinding of study

coordinator (\_4\_egb and \_10\_plansoins forms unlinked to study ID), and stored in .dta format for further management within Stata.







| SOP Plan d'analys | se statistique | |
|-------------------------|----------------|-----------------|
| SOP CRC-CHUV DM201 AN01 | | |
| SOP AGE3 DM A | N01 | Version : V01 |
| Création : | Yolanda Mülle | er / 29.11.2018 |
| Révision : | : | |
| Approbation: | IL, NS | |

The study coordinator performs monthly data monitoring. These data extracts are stored in a securised folder on the Policlinique Médicale Universitaire's server until the final analysis is completed.

The study coordinator analyses the data on a monthly basis, to identify missing items or discrepancies. If these are not, an electronic query is made in secuTrial to the person responsible of data entry for this section, who will see it and try to resolve it the next time the database in entered. Paper-based queries will be used for FP using paper data collection.

Source data validation (when applicable) is performed by the study assistant during his/her annual visits to each practice ("review A"). These visits are also an opportunity to solve all remaining queries. A final data validation takes place when data entry is considered complete. The database will be locked after all study data have been validated and monitoring review has been completed.

Data recoding:

- Removal of "test patients" from the dataset (patients created while training study physicians in using the secutrial, ID terminating by 00).
- Recoding of dates in Stata date formats (saved as strings in initial extracts)
- Treatments: manual review of treatment without ATC-code, for data entry mistakes or items missing in the predefined treatment list

# Data versioning and naming:

- Raw data extracts are saved every month in the "Raw" folder, sub-folder with the extraction date
- Recoded data are saved every month in the "Rec" folder, sub-folder with the extraction date
- At the end of data collection, a final dataset will be extracted and used for final analysis.

#### Metadata:

Project level: Identifier:

Creator: Yolanda Müller Chabloz

Affiliation: Department for ambulatory Care and Community Medicine – University of Lausanne –

Title: Active Geriatric Evaluation program – AGE4: Implementation of an electronic comprehensive assessment and management tool for geriatric syndromes in family medicine

Date: 2018 - 2021 Language: french

Funder: Swiss National Fund

HostingInstitution: Department for ambulatory Care and Community Medicine - University of

Lausanne - Switzerland

["Readme" file to be developped]

In addition to the study-specific variables, the following information is associated with each data export:

cn/casenodes: Table de base avec une ligne par patient

- mnppid : Identifiant patient secuTrial permettant de lier avec les autres tables.
- (Add-ID) mnpaid : Identifiant du sujet.

(Centre information) ctr/centres: Table des centres

(Queries and Comments) cts/comments & qas/queries : tables des commentaires et requêtes.

- ffcolname : Nom de la variable associée
- qacdate : Date du commentaire/requête
- gaccontent : Contenu du commentaire/requête.







| SOP Plan d'analys | e statistique | |
|-------------------------|---------------|-----------------|
| SOP CRC-CHUV DM201 AN01 | | |
| SOP AGE3 DM AN | NO1 | Version : V01 |
| Création : Yolanda M | | er / 29.11.2018 |
| Révision : | | |
| Approbation: | II NS | |

#### (Project Setup)

1. vp/visit plan : Liste des visites (visitid + label)

2. vpfs/visitplan forms : Relation entre visite et formulaire (visitid + formid)

3. fs/forms : Liste des formulaires et sous-formulaires associés (formid + tablename + name)

4. qs/questions : Liste des groupes d'items (séparé par ligne blanche sur l'interface)

5. is/items : Liste des variable avec le libellé associé (colname + label)

\_xxx : tables associées à chaque formulaire

• mnppid : Identifiant patient

• mnpdocid : Identifiant de l'enregistrement.

mnpvisid : Identifiant de la visite

mnpvisno : Numéro de la visite

• mnpvispdt : Date de la visite

mnpvisfdt : Date de la première saisie de donnée

e xxx: tables associées aux sous-formulaires

mnppid : Identifiant patient

• mnpdocid : Identifiant de l'enregistrement (pour lier à la table mère)

position : Numéro de répétition-1

#### Data access

- The AGE3 secutrial database is accessed via an internet browser. Each user has a specific user name and login allowing access to different sections of the data. For example, contact information is only available to the study staff that needs to contact the patients.

- Data are crypted for transfer.

- Data are stored on the server of the CHUV, Lausanne (for storage and back-up specificaiton, see 3.1).

- Data extracts are stored on the NAS-CHUV.

- Access to different parts of the data on the NAS are also defined according to different user rights.

## Data ownership

The dataset is propriety of the University Institute of Family Medicine of the Department of Ambulatory Care and Community Medicine, University of Lausanne.

Deidentified data will be shared under a creative common CCBY license.

#### Data storage

Secutrial data are stored by the Service d'Informatique of the CHUV, Lausanne (DSI-CHUV), who is responsible data storage and back-up system.

During data collection, monthly raw extracts are saved by the data manager on the server of the Department of Ambulatory Care and Community Medicine, University of Lausanne

2 copies of the data are stored in two separate locations by the DSI CHUV.

#### Data archiving

The final recoded dataset will be stored in .csv format on the server of the Department of Ambulatory Care and Community Medicine, University of Lausanne.

Other essential documents including anonymous screening logs will be stored in pdf format on the server of the Department of Ambulatory Care and Community Medicine, University of Lausanne

Nominative inclusion logs will be stored as paper format and stored in the ISF, but electronic forms will be destroyed.







| SOP Plan d'analyse statistique | | |
|--------------------------------|--------------------------|---------------|
| SOP CRC-CHUV DM201 AN01 | | |
| SOP AGE3 DM A | N01 | Version : V01 |
| Création : | Création : Yolanda Mülle | |
| Révision : | | |
| Approbation: | IL, NS | |

All contact information will be destroyed at the end of data collection.

All study data will be archived for a minimum of 10 years after study termination or premature termination of the clinical trial. Electronic data will be stored at the Lausanne University Hospital server.

Paper study data (apart from source medical files which will remain in the FP's practice and stored according to specific regulation) will be stored at the Policlinique Médicale Universitaire in Lausanne for a period of ten years under the responsibility of the principal investigator.

## Access to data for analysis:

- Study statistician (Isabella Locatelli): access to raw and recoded data
- Study coordinator (Yolanda Müller): access to recoded data

Parts of the recoded data will be shared with partners for the following subanalyses: Polymedication:

- 6. Processus + 12. Traitement + 3. Inclusion shared with medical student working on polymedication
- Recoded and anonymised data (containing patient study ID, medication, and coded diagnosis) will be shared with the Pharmacy staff of the HUG (Geneva University Hospital) for running the PIM-check tool (automated analysis of inappropriate medication) Economic analysis
- Access to recoded data will be given to Clémence Perraudin, health economist at the Department of Ambulatory Care and Community Medicine, and used for the costing of the intervention

Qualitative evaluation

- Access to sociologist (Joëlle Schwarz) and physician (Ophélie Viret) in charge of qualitative evaluation of the AGE tool

#### Data sharing

Published data will be made available in a non-for-profit repository such as Zenodo after publication

There are limitations on data sharing in order to protect human personal data.

Prof. Senn will decide when to publish and if it is possible to make Research Data accompanying the article publicly available including whether to supply research data to a new user.

Data deidentification will be conducted by a data manager to make anonymized datasets publicly available.

## In particular:

- Physician and patient ID will be recoded
- Location will be discarded (canton, CMS)
- Date of birth replaced by age in years at inclusion
- All dates referring to a specific patient will be shifted by a random number of days (consultation dates, hospitalization date, etc)
- Removal of free text fields (comments, details on profession)
- SAE information

#### Softwares for data analysis

- Stata 15.1 (College Station, USA)
- F
- MaxQDA for qualitative analysis







| SOP Plan d'analy | /se statistique | |
|-------------------------|-----------------|-----------------|
| SOP CRC-CHUV DM201 AN01 | | |
| SOP AGE3 DM A | N01 | Version : V01 |
| Création : | Yolanda Mülle | er / 29.11.2018 |
| Révision : | | |
| Approbation: | IL, NS | |

#### 7.2.1.1 Missing Data

As recommended for pragmatic trials (and nowadays for clinical trials in general), we shall follow an Intention-to-treat approach. However, we shall face the problem of a high number of missing outcome data, considering that many patients approach end-of-life age.

#### Main outcome - ADL

Missing outcome data are expected to occur mainly because of death considering the age of participants, and because of consent withdrawal (patients refusing to answer phone questionnaire). Missing outcome date cannot be considered missing completely at random, as patients approaching end-of-life, usually with a worse functional status, are more likely to refuse to answer the questionnaire. However, ADL may be imputed (assuming a Missing at random MAR mechanism) using following covariates: age, sex, ADL and IADL at baseline (and at 1 year if available), schooling, previous profession, living alone, using home-based care, frequency of contact with children and "proches aidants", driving, intervention arm and GP random intercept.

We shall start by doing a complete case analyses, completed by the following simple imputations:

- Patients who died before end-of-follow-up are considered to have declined functionally
- Patients who are institutionalized before the end of the study and who withdrew (without measured outcome) are considered to have declined functionally

## Sensitivity analyses

- Last observation carried forward: ADL result at 1 year carried forward to 2 years if missing and patient not dead
- Worst-case scenario: all missing cases considered as having lost at least one ADL
- Best-case scenario: all missing outcome considered as having maintained ADL
- Multiple imputation of ADL data, based on baseline and 1-year values, age, sex, schooling, previous profession, living alone, using home-based care, frequency of contact with children and "proches aidants", driving, intervention arm and GP random intercept

#### Main outcome - WHOQOL-OLD

Partly missing WHOQOL:

As recommended by the guidelines for scoring WHOQOL, if one of the items of a specific domain is missing, a domain score should be calculated by substituting a person specific average across the completed items in the same scale. If two or more items are coded missing in these two domains, the domain score should not be calculated.

## Completely missing WHOQOL:

- If the patient died, we shall considered his score to be 0 (standardised scale).
- Multiple imputation of WHOQOL-score, using baseline and 1-year values, age, sex, schooling, previous profession, living alone, using home-based care, frequency of contact with children and "proches aidants", driving, intervention arm and GP random intercept

#### Other outcomes

For time to event analysis (time to institutionalization, time to death), drop-outs will be censored. If date of end of follow-up is missing, we shall randomly select date between last consultation recorded and date of reported end of follow-up.







| SOP Plan d'ana | lyse statistiq | ue |
|---------------------|----------------|---------------------|
| SOP CRC-CH | IUV DM20 | )1 AN01 |
| Création : | Yolanda | Müller / 29.11.2018 |
| Révision : | | |
| Approbation: IL, NS | | |

Otherwise, we expect that missing data among the planned adjustment factors will be limited. Multiple imputation is therefore not planned for additional variables.

We do not expect major missingness in variables collected as part of the medical file. Some events may not be recorded in the medical file and will not be captured by our data collection, but we have no ways of correcting this. Process data might be more difficult to obtain in the control group because of less attention given to file notes, resulting in a higher number of missing data. This will be checked in the interim analysis.

## 7.2.1.2 Extreme values

Predefined checks included in the data collection software prevented a number of aberrant values. For the main outcomes, model post-estimation will include assessment of outliers, which may be excluded on a case-by-case assessment.

## 7.2.2 Descriptive analyses

## 7.2.2.1. Data cleaning

Data monitoring will be done continuously (at least monthly) by the study coordinator, blinded to group allocation. BAT data will be monitored separately, after unlinking of the data with patient and FP identifier.

7.2.2.2. Descriptive analysis

For continuous variables: mean, standard deviation, interquartile range, min/max and boxplot, per arm For ordinal variables: median, interquartile range, mode, min/max and bar plot, per arm For categorical variables: Cross-tabulation, per arm

7.2.2.3. Demographical characteristics

Basic sociodemographic and clinical characteristics (comorbidities) of patients and FP characteristics will be described for both arms.

Patient characteristics will also be compared by sex/gender.

## 7.2.3 Multivariate analyses

Hypothesis 1.1

The primary analysis will compare the difference in proportion of patients having lost at least 1 IADL after 2 years between intervention and control group, using a generalised 2-level linear mixed model with a logit distribution. Clustering by FP will be taken into account by the mixed model ("physician effect"). Baseline and 1-year IADL will be included in the model if available (repeated measures). Important determinants of FP variance will be explored and included in the model if relevant (practice size and type, age, gender of FP, specialty type, comprehensiveness of care)

The following analyses are also planned to be performed by the study statistician after database closure:

- Difference in proportion of patients having lost at least 1 ADL after 2 years between intervention and control group, using a generalised linear mixed model
- Difference in WHOQOL-OLD after 2 years between intervention and control group, using a generalised linear mixed model







| SOP Plan d'analyse statistique | | |
|--------------------------------|--------|----------------|
| SOP CRC-CHUV DM201 AN01 | | |
| SOP AGE3 DM AN | N01 | Version : V01 |
| Création : Yolanda Mül | | r / 29.11.2018 |
| Révision : | | |
| Approbation: | IL, NS | |

 Difference in IADL, ADL and WHOQOL-OLD difference (delta) between baseline measurement and after 2 years between intervention and control group, using a generalised linear mixed model

For the primary outcome, subgroup analysis will be performed by patient characteristics (gender, age category, baseline disability, comorbidities) and FP characteristics (gender, age, urban/rural/semi-urban)

- Number of hospital admissions, institutionalizations, emergency visits and routine visits using a linear mixed model
- Survival analysis of time to institutionalization and time to death

For process evaluation, the number of geriatric syndromes suspected, confirmed and acted upon will be compared after 2 years. Implementation of management strategies (investigations, medication adaptation, referral to specialty care, supportive measures) included in AGE will be compared between both groups, based on the information in the medical file. Based on a predefined scale, FP adhesion to the AGE tool will be estimated for each patient.

Sensitivity analyses

We will also whether the primary outcome is dependent of the % adhesion to AGE.A complier average causal effect analysis will be used to estimate the effect of the intervention in the intervention group, had all FPs adhered to it[15, 16].

A more classical "per protocol" analysis will restrict the analysis to the population of patients in the intervention group which had both BAT performed (at least 7 out of 8 items screened) in the planned timeframe, and at least 50% adherence of FP to the AGE tool.

#### Qualitative analysis

A thematic analysis will be performed throughout the data collection using MaxQDA. A first code system will be derived from the response to research questions. After review of the material by the first coder, the material will be coded again independently by a second researcher and results will be compared in order to ensure coding consistency (cross-checking procedure). Codes will be encompassed in themes with a broader level of meaning and organized in a way that answers the research questions.







| SOP Plan d'ana | yse statistiq | ue |
|---------------------|---------------|---------------------|
| SOP CRC-CH | HUV DM20 | 1 AN01 |
| Création : | Yolanda I | Müller / 29.11.2018 |
| Révision : | | |
| Approbation: IL, NS | | |

## 8. REFERENCES

- 1. Rosso AL, Eaton CB, Wallace R, Gold R, Stefanick ML, Ockene JK, Curb JD, Michael YL: Geriatric syndromes and incident disability in older women: results from the women's health initiative observational study. *Journal of the American Geriatrics Society* 2013, 61(3):371-379.
- 2. Gill TM, Baker DI, Gottschalk M, Peduzzi PN, Allore H, Byers A: A Program to Prevent Functional Decline in Physically Frail, Elderly Persons Who Live at Home. New England Journal of Medicine 2002, 347(14):1068-1074.
- Lawton MP, Casten R, Parmelee PA, Van Haitsma K, Corn J, Kleban MH: **Psychometric characteristics of the minimum data set II: validity**. *Journal of the American Geriatrics Society* 1998, **46**(6):736-744.
- 4. Katz S: Assessing self-maintenance: activities of daily living, mobility, and instrumental activities of daily living. *Journal of the American Geriatrics Society* 1983, **31**(12):721-727.
- 5. Spector WD, Fleishman JA: Combining activities of daily living with instrumental activities of daily living to measure functional disability. The journals of gerontology Series B, Psychological sciences and social sciences 1998, 53(1):S46-57.
- 6. Dalby DM, Sellors JW, Fraser FD, Fraser C, van Ineveld CH, Pickard L, Howard M: Screening seniors for risk of functional decline: results of a survey in family practice. Canadian journal of public health = Revue canadienne de sante publique 1999, 90(2):133-137
- 7. Ciesla JR, Shi L, Stoskopf CH, Samuels ME: Reliability of Katz's Activities of Daily Living Scale when used in telephone interviews. Eval Health Prof 1993, 16(2):190-203.
- 8. Hopman-Rock M, van Hirtum H, de Vreede P, Freiberger E: Activities of daily living in older community-dwelling persons: a systematic review of psychometric properties of instruments. Aging Clin Exp Res 2018.
- 9. Leplège A, Perret-Guillaume C, Ecosse E, Hervy MP, Ankri J, von Steinbüchel N: **Un nouvel** instrument destiné à mesurer la qualité de vie des personnes âgées : le WHOQOL-OLD version française. La Revue de Médecine Interne 2013, **34**(2):78-84.
- 10. Power M, Quinn K, Schmidt S: **Development of the WHOQOL-Old Module**. *Quality of Life Research* 2005, **14**(10):2197-2214.
- 11. Joanovic E, Kisvetrova H, Nemcek D, Kurkova P, Svejdikova B, Zapletalova J, Yamada Y: Gender differences in improvement of older-person-specific quality of life after hearing-aid fitting. Disability and health journal 2018.
- 12. Romero PS, de Souza EN, Rodrigues J, Moraes MA: Changes in quality of life associated with surgical risk in elderly patients undergoing cardiac surgery. International journal of nursing practice 2015, 21(5):592-597.
- 13. Volter C, Gotze L, Dazert S, Falkenstein M, Thomas JP: Can cochlear implantation improve neurocognition in the aging population? *Clinical interventions in aging* 2018, 13:701-712.
- 14. Yamada Y, Svejdikova B, Kisvetrova H: Improvement of older-person-specific QOL after hearing aid fitting and its relation to social interaction. *Journal of communication disorders* 2017, **67**:14-21.
- 15. Fairhall N, Sherrington C, Cameron ID, Kurrle SE, Lord SR, Lockwood K, Herbert RD: A multifactorial intervention for frail older people is more than twice as effective among those who are compliant: complier average causal effect analysis of a randomised trial. *Journal of physiotherapy* 2017, 63(1):40-44.
- 16. Peugh JL, Strotman D, McGrady M, Rausch J, Kashikar-Zuck S: **Beyond intent to treat** (ITT): A complier average causal effect (CACE) estimation primer. *Journal of school psychology* 2017, **60**:7-24.